CLINICAL TRIAL: NCT03179449
Title: MR Imaging of Inflammatory Responses in the Central Nervous System With Ferumoxytol-Enhanced MRI (Pediatric Brain Tumor Protocol)
Brief Title: In Vivo Characterization of Macrophages in Pediatric Patients With Malignant Brain Tumors Using Ferumoxytol-enhanced MRI
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Accrual Factor
Sponsor: Michael Iv (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Michael Iv, Clinical Assistant Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-39245; NCI-2017-00959 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PEDSBRNCNS0008 (Other: Stanford Cancer Institute); P30CA124435 (NIH); PEDSBRNCNS0008 (Other: OnCore)
Record Dates: First submitted 2017-06-05; First posted 2017-06-07 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Childhood Brain Neoplasm
MeSH Terms: interventions — Diagnosis; Dynamic Contrast Enhanced Magnetic Resonance Imaging; Surgical Procedures, Operative; Ferrosoferric Oxide; Tissue Array Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (ferumoxytol-enhanced MRI) (Experimental): All subjects in the experimental arm will have a single intravenous dose of ferumoxytol (5 mg Fe/kg), to be administered 24 hours before the subject undergoes ferumoxytol-enhanced magnetic resonance imaging (MRI). These subjects will subsequently undergo surgery, and tissue analysis of surgically resected samples (specifically the number of iron-containing and non-iron-containing macrophages) will be correlated with imaging features on ferumoxytol-enhanced MRI.
  Interventions: Diagnostic Test: Diagnostic (ferumoxytol-enhanced MRI); Procedure: Surgery; Drug: Ferumoxytol; Other: Tissue Analysis

INTERVENTIONS:
Diagnostic Test: Diagnostic (ferumoxytol-enhanced MRI) — Undergo ferumoxytol-enhanced MRI
  Other Names: CONTRAST ENHANCED MRI; Contrast-enhanced MRI
Procedure: Surgery — Undergo surgical resection
Drug: Ferumoxytol — Given IV
  Other Names: Feraheme; FERUMOXYTOL NON-STOICHIOMETRIC MAGNETITE
Other: Tissue Analysis — Correlative analysis for macrophage detection and quantification. This applies for all patients in the experimental arm who undergo ferumoxytol infusion.

SUMMARY:
This pilot early phase I trial studies how well ferumoxytol-enhanced magnetic resonance imaging (MRI) correlates with inflammatory (macrophage) responses in pediatric patients with malignant brain tumors. If there is good correlation, ferumoxytol-enhanced MRI can serve as a noninvasive imaging biomarker of inflammation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To establish the magnetic resonance (MR) imaging signal characteristics of macrophages in pediatric patients (>= 2 years old) with newly diagnosed malignant brain tumors using ferumoxytol, an ultrasmall superparamagnetic iron oxide (USPIO) particle.

SECONDARY OBJECTIVES:

I. To correlate the MRI signal of ferumoxytol uptake in macrophages with the number of macrophages in surgical tumor specimen at histopathology.

OUTLINE:

Patients receive a single intravenous infusion of ferumoxytol over 15 minutes. After 24 hours, patients undergo ferumoxytol-enhanced magnetic resonance imaging (MRI). Patients will then undergo MRI-localized tissue sampling and tumor resection.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with suspected malignant brain tumor on diagnostic MR imaging who will undergo a resection

Exclusion Criteria:

* Informed consent cannot be obtained either from the patient or legal representative
* Severe coexisting or terminal systemic disease that may interfere with the conduct of the study
* Contraindication to MRI (metal implants)
* Hemosiderosis/hemochromatosis
* Iron overload from any cause (not just hemosiderosis or hemochromatosis), even if secondary to frequent blood transfusions, severe chronic hemolysis, excess dietary or parenteral iron, or any other etiology
* Known hypersensitivity to ferumoxytol or any of its components
* Pregnant patients

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Iron concentration measurements | Day 1
  Obtain susceptibility measurements and relaxation times (R2, R2*, R2') in patients receiving ferumoxytol.

SECONDARY OUTCOMES:
Macrophages on histopathology | Days 2-4
  Determine the number of macrophages in tissue samples at histopathology.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Iv, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No